CLINICAL TRIAL: NCT03072862
Title: Cochlear Implant and Healthy Aging: A Multinational, Multicentre Observational Study
Brief Title: Evaluation of the Benefits for Overall Health Following Cochlear Implant Treatment in the Elderly Population
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL5671
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Hearing Loss
Keywords: Cochlear implant treatment, aging adults
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Commercial Nucleus Cochlear Implant Systems
  Interventions: Device: Commercial Nucleus Cochlear Implant Systems

INTERVENTIONS:
Device: Commercial Nucleus Cochlear Implant Systems — Commercially available Nucleus Cochlear Implant Systems, including Data Logging functionality

SUMMARY:
The purpose of this study is to show that cochlear implant treatment improves the overall health related quality of life and general well-being in elderly individuals.

DETAILED DESCRIPTION:
The study is designed as an observational prospective repeated measures study with each subject acting as his/her own control. Subjects are evaluated subjectively at pre- and post-operative intervals that coincide with their routine visits to the clinic. Outcomes from routine practice and application of cochlear implant intervention are recorded through observational measures using clinical standards scales used widely in geriatrics and audiology. The study is aimed at collection of data for patients who have already made the decision together with their implant centre clinician for an implant device from the company Cochlear. Patients are approached for study participation prior to surgery by the caring clinician on a consecutive and voluntary basis and on condition of signing the patient informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral CI candidates with bilateral post-lingual deafness with intention to treat
* ≥ 60 years at first unilateral cochlear implant
* Implant ear: meets all local criteria for cochlear implant treatment
* Contralateral ear: average pure tone thresholds indicate a moderately-severe to profound hearing loss (4 freq. average: 0.5, 1, 2 and 3 or 4 kHz > 56 dBHL).
* Willingness to participate in and to comply with all study procedures
* Fluency in languages used to assess clinical performance
* Appropriate expectations from routine cochlear implant treatment
* Able to decide on study participation personally and independently sign their consent

Exclusion Criteria:

* Significantly/severely dependent or fragile
* Unable to provide consent personally
* Unable to complete questionnaires for self-assessment independently
* Unilateral hearing loss
* Sequential and simultaneous bilateral cochlear implant recipients
* Ossification or other cochlear anomalies preventing full electrode insertion
* Retro cochlear or central origins of hearing impairment.
* Significant comorbidities preventing study participation (e.g. blindness, immobility or in a wheel chair, severe aphasia)
* Medical contraindications to surgery
* Clinic Standard fail criteria for cochlear implant candidacy in regards to chronic depression, dementia, and cognitive disorders.
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly routine clinical patients with permanent hearing loss seeking treatment with a commercial cochlear implant system.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, PhD, Study Director — Cochlear
Locations (8):
- France (2):
  - Groupe Hospitalier de La Pitié Salpétrière, Paris
  - ENT Department-Hôpital Purpan, Toulouse
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center (Beilinson), Petah Tikva
- Italy (2):
  - ENT Otosurgery Department-Azienda Ospedaliera di Padova, Padua
  - ENT Department Ospedale Guglielmo da Saliceto, Piacenza
- Spain (2):
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Clinica Universitaria de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuda D, Manrique M, Ramos A, Marx M, Bovo R, Khnifes R, Hilly O, Belmin J, Stripeikyte G, Graham PL, James CJ, Greenham PV, Mosnier I. Improving quality of life in the elderly: hearing loss treatment with cochlear implants. BMC Geriatr. 2024 Jan 4;24(1):16. doi: 10.1186/s12877-023-04642-2. PMID 38178036
- [Derived] Marx M, Mosnier I, Belmin J, Wyss J, Coudert-Koall C, Ramos A, Manrique Huarte R, Khnifes R, Hilly O, Martini A, Cuda D. Healthy aging in elderly cochlear implant recipients: a multinational observational study. BMC Geriatr. 2020 Jul 23;20(1):252. doi: 10.1186/s12877-020-01628-2. PMID 32703167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants were recruited in 8 centres from 06 November 2017 to 21 March 2022.
Period: Overall Study
Arm/Group | Commercial Nucleus Cochlear Implant Systems
Started | 100
Completed | 82
Not Completed | 18
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 4
Not completed — Physician Decision | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 2 participants did not meet the inclusion/exclusion criteria and were excluded from analysis.
Arm/Group | Commercial Nucleus Cochlear Implant Systems
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 35
  Israel | 7
  France | 35
  Spain | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Health Related Quality of Life Following Cochlear Implant Treatment
Description: Assessed via the Health Utilities Index Mark III (HUI 3) questionnaire. HUI-3 classification system consists of 8 attributes including vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain. HUI-3 values range from -0.36 to 1.00. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change in scores is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: pre-implant surgery, 12 months post-surgery
Population: Data were available for 85 participants for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Commercial Nucleus Cochlear Implant Systems
Number analyzed (Participants) | 85
units on a scale
  Multi-attribute score | 0.14 [0.08 to 0.19]
  Hearing single-attribute | 0.22 [0.16 to 0.29]
  Speech single-attribute | 0.08 [0.03 to 0.12]

2. Primary Outcome: Change in Health Related Quality of Life Following Cochlear Implant Treatment
Description: Assessed via the Health Utilities Index Mark III (HUI 3) questionnaire. HUI-3 classification system consists of 8 attributes including vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain. HUI-3 values range from -0.36 to 1.00. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change in scores will be presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: pre-implant surgery, 18 months post-surgery
Population: Data were available for 82 participants for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Commercial Nucleus Cochlear Implant Systems
Number analyzed (Participants) | 82
units on a scale
  Multi-attribute | 0.13 [0.07 to 0.18]
  Hearing single-attribute | 0.25 [0.18 to 0.31]
  Speech single-attribute | 0.08 [0.03 to 0.14]

ADVERSE EVENTS:
Time Frame: 20 months
Description: Incidents defined as "any malfunction or deterioration in the characteristics or performance of a device made available on the market, including use-error due to ergonomic features, any inadequacy in the information supplied by the manufacturer as well as any undesirable side-effect" were collected. One participant died; the cause of death was not related to the device.
Arm/Group | Commercial Nucleus Cochlear Implant Systems
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Commercial Nucleus Cochlear Implant Systems (N=100)
Magnet dislocation after MRI (Magnetic Resonance Imaging) (Product Issues) | 2 (100)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to generate at least two joint publications by the clinical investigator(s), with support from the sponsor using collective data. Publications are requested to be reviewed by the sponsor at least 30 days in advance to submission for publication.

Investigators are able to publish their local data separately. The sponsor kindly requests a copy of manuscripts intended for submission for publication least 60 days in advance of submission.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03072862/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03072862/SAP_001.pdf